

## Believing is Seeing

840 Walnut Street Philadelphia, PA 19107 215-928-3000 1-877-AT-WILLS www.willseye.org

visuALL Validation Study 1.2 Principal Investigator: M. Reza Razeghinejad, MD

> NCT03804684 IRB# 18-768E

Study Protocol November 6, 2018



## visuALL Validation Study 1.2

| Protocol Number | 001 |
|---|---|
| Principal Investigator (PI) | M. Reza Razeghinejad MD |
| PI email | mrazeghi@willseye.org |
| Coordinating Center | Wills Eye Hospital; 840 Walnut Street, Philadelphia, PA 19107 |
| Protocol Version | 1.2 |
| Date | October 1, 2018; rev. November 6, 2018 |
| Protocol Authors | L. Jay Katz, MD |
| | Dr. Alberto Gonzalez Garcia |
| Liaison/Olleyes | Dr. Alberto Gonzalez Garcia |
| | gonzalezao@olleyes.com |
| Sponsor | Olleyes, Inc. |
| | 11 Hillcrest Dr, Randolph |
| | NJ 07869 |
| | 973-567-8068 |



| Study Objective To determine age-adjusted reference values of the visuALL Field Analyze (vFA), to assess the repeatability for each parameter and correlate them with a Standard Automatic Perimetry (SAP) parameters. Study Rationale Standard Automatic Perimetry (SAP) is the gold standard test for the evaluation of different diseases of the visual pathway like glaucoma. Its main goal is to measure the differential light sensitivity at several locations of the central field of vision. Nevertheless, the accuracy of the |
|---|
| with a Standard Automatic Perimetry (SAP) parameters. Study Rationale Standard Automatic Perimetry (SAP) is the gold standard test for the evaluation of different diseases of the visual pathway like glaucoma. Its main goal is to measure the differential light sensitivity at several |
| Study Rationale Standard Automatic Perimetry (SAP) is the gold standard test for the evaluation of different diseases of the visual pathway like glaucoma. Its main goal is to measure the differential light sensitivity at several |
| evaluation of different diseases of the visual pathway like glaucoma. Its main goal is to measure the differential light sensitivity at several |
| main goal is to measure the differential light sensitivity at several |
| locations of the central field of vision. Nevertheless, the accuracy of the |
| current device is limited by several factors like the inherent inconsistence |
| of the psychophysical test, stressful examinations and frequency of |
| testing among others. <sup>1,2</sup> |
| Several devices have been developed since the advent of the Octopus |
| Perimeter <sup>3-5</sup> and the Humphrey Field Analyzer (HFA), <sup>6,7</sup> in an effort to |
| improve the early detection glaucoma. <sup>8,9</sup> Examples of these visual field |
| test variants are implemented using laptops and iPads and virtual reality |
| headsets. <sup>10-13</sup> |
| These modalities bring portability but the lack of fixation methods, |
| environmental control and hardware standardization may limit its wide |
| usage. |
| The main goal of this study is to evaluate the repeatability of a novel |
| psychophysical platform that takes advantage of a Head Mounted Devic |
| (HMD) with eye tracking capabilities. Other objectives of this study |
| include the development of an initial reference database and the |
| evaluation of its correlation with HFA parameters. |

| Study Design | visuALL-1 is a cross-sectional observational study. The primary endpoint |
|---|---|
| | of the study will be at end of the recruitment phase. |
| Participants | A group of healthy subjects and patients with glaucoma; between 21 and |
| | 80 years old will be invited to participate in the study. A total of 50 |
| | healthy eyes and an additional 50 eyes with glaucoma will be recruited |
| | for this study. |
| | All subjects will undergo a complete ophthalmologic examination at the |
| | glaucoma department of Wills Eye Hospital. Each examination will |
| | include refraction, slit lamp biomicroscopy of the anterior segment, IOP |
| | measurement, BCVA, visual field and visuALL Field Analyzer (vFA) testing, |
| | gonioscopy and dilated stereoscopic fundus examination of the retina |
| | and optic nerve head. Data about family history of glaucoma will also be |
| | recorded. |



| | Study Groups: | |
|---|---|---|
| | Study Groups: 1. Control group: Healthy eyes (n=50) | |
| | 1. Control group: Healthy eyes (n=50) | |
| | 2. Glaucoma group: Chronic Open Angle Glaucoma (COAG) eyes | |
| | (n=50) | |
| | - 30 eyes with mild COAG | |
| | - 20 eyes with moderate COAG | |
| | The recruitment process of healthy subjects will include a stratification | |
| | based on age as indicated in the table below. | |
| | Age Group (years) | Eyes |
| | 30 - 39 | 10 |
| | 40 - 49 | 10 |
| | 50 - 59 | 10 |
| | 60 - 69 10 | |
| | 70 and more 10 | |
| | Individuals of different races will be included but no single ethnic group | |
| | will encompass more than 50%. 15% of gender differences will be | |
| | allowed. | |
| | The clinical study plan will be reviewed and approved by Wills Eye | |
| | Hospital Institutional Review Board (IRB). | |
| Healthy criteria | Normal appearing optic nerve and retina | |
| , | • IOP < 19 mmHg. | |
| | <ul> <li>Normal SAP results in both eye</li> </ul> | s (See SAP criteria) |
| COAG criteria | , | c nerve and/or retina (i.e. increased |
| COAG CITIEITA | | |
| | | inning or RNFL defects indicative of |
| | glaucoma) | /C CAD :: ` ` |
| | Abnormal SAP results in the stu | |
| Exclusion criteria | 1. A spherical refraction outside ± | : 3.0 D and cylinder correction |
| | outside 2.0 D. | |
| | , | fixation losses and false negatives |
| | >25% and/or observable testing | , |
| | 3. Unreliable vFA (>25% false pos | , , |
| | 4. SAP abnormality with a pattern | of loss which is consistent with a |
| | neurologic and/or other ocular | diseases than glaucoma. |



| | 5. Intraocular surgery in the study eye (except non-complicated |
|---|---|
| | cataract or refractive surgery performed more than 6 months |
| | before enrollment and without posterior capsule opacification). |
| | 6. History of systemic condition known to affect visual function. |
| | 7. History of medication known to affect visual function. |
| Instrumentation | 1. Refraction (autorefractor) |
| | 2. Tonometry (Goldmann) |
| | 3. SAP Humphrey Field Analyzer (HFA) 24-2, Swedish Interactive |
| | Threshold Algorithm (SITA) Standard Strategy (Carl Zeiss Meditec, |
| | Inc. Dublin, CA) (single session). |
| | 4. visuALL <i>Pro</i> (Olleyes, Inc. Randolph, NJ) (single session). |
| Within Normal | Pattern Standard Deviation significant within 95% normal limits, |
| Limits SAP criteria | Glaucoma Hemifield test within normal limits, and no other pattern of |
| | loss which is consistent with a neurologic and/or ocular disease. |
| vFA reliability | False positives, fixation losses and false negatives >25% and/or |
| criteria | observable testing artifacts |
| vFA Description | vFA <i>Pro</i> will be used for this validation study. The visuALL system is |
| | composed of two main parts - the hardware and the software. |
| | The hardware includes three main components: A Head Mounted Device |
| | (HMD) also known as Virtual Reality (VR) headset, a Laptop and a |
| | Bluetooth connected handpiece. |
| | The HMD is powered by FOVE (Fove, Inc. Tokyo, Japan). This HMD weight |
| | 520g and includes a Wide Quad High Definition Organic Light Emitted |
| | Diode (WQHD OLED) display with a resolution of 2560x1440 pixels with a |
| | refresh rate pf 70Hz. The display is divided in two halves (one for each |
| | eye) with a resultant resolution of 1280x1440 pixels on each half. The |
| | display measures 125.4 x 70.56 mm and it is placed at a distance to |
| | subtend a field of view (FOV) up to 100 degrees. |
| | The HMD includes several tracking systems, inertial measurement units |
| | (IMUs) consisting of gyroscopes and accelerometers, in addition to |
| | infrared-based (IR) position tracking with two arrays of 6 IR sensors. |
| | The HMD uses 2 eye-tracking system including infrared cameras with a |
| | frame rate of 120fps. The eye-tracking system has a resolution of less |
| | than 1 degree. |
| | The main PC components are a graphic processing units (GPU) NVIDIA |
| | GeForce GTX 970, a central processing unit (CPU) Intel Core i7 7th Gen |
| | 7820HK (2.90 GHz), random access memory (RAM) of 32GB, a hard disk |



| | T | ( | | 1 = 6 | |
|---|---|---|---|---|---|
| | drive (HDD) of 1 TB and 3 main interfaces: one High Definition Media | | | | |
| | Interface (HDMI), one Universal Serial Bus (USB) 3.0 and two USB 2.0. | | | | |
| | The PC runs and Operating System (OS) WINDOWS 10 64-bit. The PC | | | | bit. The PC |
| | networking protocols are Killer Ethernet E2400 10/100/1000 Gigabit | | | | 00 Gigabit |
| | Ethernet LAN (RJ-45 port), Wi-Fi Dual-Band (WLAN) 2.4GHz and 5GHz and Bluetooth 4.1 | | | | z and 5GHz |
| | | The visuALL software includes three main testing protocols. | | | |
| | | neters | SupraT | NormalT | FlickerT |
| | | e (degrees) | 24 | 24 | 24 |
| | | ground Illumination (cd/m²) | 10 | 10 | 50 |
| | | lus Locations | 54 | 54 | 54 |
| | Stimu | lus Size (degrees) | 0.43 | 0.43 | 5 |
| | Stimu | lus Duration (ms) | 150 | 150 | Up to 200 |
| | Stimu | lus Intensity (cd s/m²) | 100 | Variable | 50 |
| | Inter- | stimulus Time (ms) | Random | Random | Random |
| | Fixatio | on Control | Eye tracking | Eye tracking with dynamic stimulation-grid | |
| | | | - T | within a threshold | |
| | | | otherwise pa | aused. Blinking co | ontrol |
| vFA Outcome | Retinal sensitivity at each location | | | | |
| Measurements | Mean retinal sensitivity at each quadrant | | | | |
| | • [ | Mean retinal sensitivity a | t each hemifi | eld | |
| | Mean retinal sensitivity | | | | |
| Analyses | | | demographic | | |
| | | References values | | | |
| | | Reliability indexes for HFA | \ and vEA var | iahles | |
| | | • | | | |
| Deferences | | Agreement between HFA | | | . : |
| References | | Heijl A, Lindgren A, Lindgı | | | |
| | | glaucomatous visual field | • | | |
| | 2. F | Russell RA, Crabb DP, Ma | lik R, Garway- | -Heath DF. The | relationship |
| | k | between variability and s | ensitivity in la | irge-scale long | itudinal visual |
| | f | field data. Invest Ophthal | mol Vis Sci. 2 | 012;53:5985-5 | 990. |
| | 3. 9 | Spahr J, Fankhauser F, Be | bié H. Advand | ces in the auto | mation of |
| | ļ | perimetry. Klin Monbl Au | genheilkd. 19 | 76;168:84-6. | |
| | | Spahr J, Fankhauser F, Jer | _ | | eriences with |
| | | the Octopus automatic po | , | · | |
| | | 1978;172:470-7. | | | |
| | | • | itomated na | imotru booka | cound |
| | | Portney GL, Krohn MA. A | · | | |
| | j | instruments and methods | s. Surv Ophth | almol. 1978;22 | 2:2/1-8. |



| | 6. Beck RW, Bergstrom TJ, Lichter PR. A clinical comparison of visual field testing with a new automated perimeter, the Humphrey Field Analyzer, and the Goldmann perimeter. Ophthalmology. 1985;92:77-82. |
|---|---|
| | 7. Brenton RS, Phelps CD. The normal visual field on the Humphrey field analyzer. Ophthalmologica. 1986;193:56-74. |
| | 8. Bosworth CF, Sample PA, Johnson CA, Weinreb RN. Cur- rent practice with standard automated perimetry. Semin Ophthalmol 2000;15:172–181. |
| | 9. Delgado MF, Nguyen NTA, Cox TA et al. Automated perimetry: a report by the American Academy of Ophthalmology. Ophthalmology 2002;12:2362–2374. |
| | 10. Wu Z, Guymer RH, Jung CJ, et al. Measurement of retinal sensitivity on tablet devices in agerelated macular degeneration. Trans Vis Sci Tech. 2015;4:13. |
| | 11. Tahir HJ, Murray IJ, Parry NRA, Aslam TM. Optimization and Assessment of Three Modern Touch Screen Tablet Computers for Clinical Vision Testing. PLoS ONE 2014;9: e95074. |
| | 12. Vingrys AJ, Healey JK, Liew S, et al. Validation of a tablet as a tangent perimeter. Trans Vis Sci Tech. 2016;5:3. |
| | 13. Prea SM, Yu Kong YXG, Mehta A, He M, Crowston JG, Gupta V, Martin KR, Vingrys AJ. Six-month Longitudinal Comparison of a |
| | Portable Tablet Perimeter With the Humphrey Field Analyzer. Am J<br>Ophthalmol 2018;190:9–16. |
| Proposed Due Date Fe | ebruary 2019 |
| for Analysis of | |
| Primary End Point | |
| Data: | |
| Planned TI | he Study will plan to submit abstracts for 2019 ARVO. Subsequently two |
| Publications & m | nanuscripts will be written and submitted to Journal of Glaucoma and |
| <b>Abstract</b> O | )phthalmology. |
| Submissions: | |